CLINICAL TRIAL: NCT05861661
Title: The Connection Between Attachment, Emotional Regulation and Mentalization Failures in Anorexia Nervosa
Brief Title: Social Cognition in Patients With Anorexia Nervosa- the Study Examines Social Understanding in Patients With AN Via Questionnaire and Computer Tasks
Status: Completed | Type: Observational
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0051-20-ZIV
Record Dates: First submitted 2020-07-12; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2020-07

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The study do not include an intervention — The study do not include an intervention

SUMMARY:
The current research has two goals: first to validate the Hebrew version of a new measurement for assessing mentalization failures. The second goal is to examine the connection between attachment, emotional regulation strategies, mentalization, and specific mentalization failures - As they manifested in anorexia nervosa (AN) compared with non-patient controls. The study includes computer tasks, questionnaires and two short tasks administrated by the examiner.

DETAILED DESCRIPTION:
Study goals:

1. To validate the Hebrew version of the Movie for the Assessment of Social Cognition (MASC) which asses mentalization ability and mentalization failures (Dziobek et al., 2006). This version of the MASC was recently designed by the study group in Haifa University. The validation of this version of the MASC will be done by comparing patients with AN to non-patients.
2. To examine the connection between attachment styles, emotional regulation strategies, mentalization, and specific mentalization failures.

Study Hypotheses:

1. In respect to the first goal of the study, we hypothesize that a. a significant correlation between the MASC and other tools examining different aspects of mentalization (RME, CAM, TAS and RFQ) will be fond; b. different patterns of mentalization will be found between the clinical group and the control group on the MASC. More specifically, patients with AN will show more hypo-mentalization tendencies on the MASC then the control group.
2. regarding the second goal of the study, we hypothesize that the connection between attachment and mentalization failures will be mediated via emotional regulation strategies. More specifically, we anticipate that the connection between avoidant attachment and hypo-mentalization will be mediated via emotional isolation strategy and the connection between anxious attachment and hyper-mentalization will be mediated via emotional flood.

Method:

Participants This study will include 120 participants at the ages of 16-26. The participants will be assigned into two groups. The AN group will include 60 women diagnosed according to the DSM-5 (APA, 2013) as suffering from AN and are currently hospitalized. The control group will include 60 women participants, which will be screened and excluded if found to be suffering from any type ED, have a psychiatric background or any chronic disease. The control group will be recruited threw Haifa university. The control group session will take place in Haifa university.

Measures

Measures of mentalization

The Movie for Assessment of Social Cognition (MASC) (Dziobek et al., 2006) - Hebrew version. This task was designed to serve as a refined, easily-administered, ecologically-valid measure of ToM and ToM errors. It was originally shown to discriminate between adults with Asperger syndrome and healthy controls, and has since been used in studies researching ToM, mentalization and mentalization deficits in different psychopathology's, including AN and SAD. It was also translated to Spanish and Norwegian, and was found to be valid in these languages (Lahera et al., 2014, Fretland et al. 2015). The task consists of a film depicting four young adults getting together for dinner. The film stops at various points to pose questions regarding the thoughts, intentions and feelings of the characters. Overall, the task includes 45 multiple-choice questions; each question has one correct answer and three distractors, which can be characterized as reflecting exceeding ToM/hypermentalization, insufficient ToM/hypomentalization and concrete answers which involve no ToM. We will use the Hebrew version of the task, which was translated and dubbed for the purpose of the current research project.

Reading the Mind in the Eyes (RME)- Revised Version (Baron-Cohen et al., 2001). This task was designed to assess the ability to recognize basic and complex emotions and ToM. It has also been found to be valid when translated into other languages (Hallerbäck et al., 2009, Prevost et al., 2014). In the current study we will use the Hebrew version translated by Milo. During the task, participants are presented with 52 photographs of eyes exhibiting basic emotions (happy, sad, afraid, surprised, disgusted, angry) (Ekman & Friesen, 1976) as well as complex emotions (interested, worried, confident, fantasizing, preoccupied, friendly and suspicious) (Baron-Cohen et al., 1997). Each picture is presented twice, and participants are asked to make a forced choice between four words naming the emotion, with only one correct answer.

The Cambridge Mindreading (CAM) Face-Voice Battery - (Golan et al., 2006). This battery examines complex emotion and mental-state recognition in both visual and auditory format. In the current study we will use only the visual task, which is comprised of silent clips of adult actors, both male and female, of different ethnicities, expressing emotions facially. Fifty faces examine recognition of 20 different complex emotions and mental states (e.g., intimate, insincere). During each trial, a clip is presented and the participants are asked which of four words best describes the emotions being displayed. There is no time limit for answering. The battery provides an overall facial emotion recognition score (max =50) as well as individual scores for each of the 20 emotions assessed (pass/fail, i.e., recognized above chance or not) and an overall number of the emotions correctly recognized (max=20). The current study will use a Hebrew version of this task which was developed by Prof. Ofer Golan, one of the designers of the original English version, alongside Prof. Lily Rothschild-Yakar.

The Toronto Alexithymia Scale (TAS-20) - (Griffith, 1998). The TAS is a 20-item self-report measure, which was developed for the assessment of alexithymia, yet can also be used to measure mentalization in relation to the self (Luyten et al., 2012). The scale has 3 factors which were confirmed in several studies (Parker, Taylor, & Bagby, 2003): (a) difficulty in identifying feelings, (b) difficulty in describing feelings to others; and (c) externally oriented thinking. The scale's internal consistency (α =.81(, and test-retest reliability (r = .77) have been established (Bagby, Taylor, & Parker, 1994), and its Hebrew version showed good internal consistency (α = 0.89; Rozenstein et al. 2011) The Reflective Functioning Questionnaire (RFQ), (Fonagy et al, 2016). The RFQ is a relatively new instrument, developed as a brief, easy-to-administer, self-report screening measure of mentalization. It originally included 46 items which the participant responded to on a 6-point scale. Factor analysis yielded two main factors, assessing Certainty (RFQ_C) and Uncertainty (RFQ_U) about the mental states of self and others. These two factors allow distinguishing between the two the main mentalization impairments, hyper-mentalization and hypo-mentalization, with high scores of certainty indicating hyper-mentalization and high scores of uncertainty reflecting hypo-mentalization; low scores on both scales indicate more genuine mentalizing. The factors were relatively distinct, invariant across clinical and non-clinical samples, had satisfactory internal consistency and test-retest stability, and were largely unrelated to demographic features. The questionnaire's developers have since designed a short, 8-item version, consisting of the highest loading items on their respective factor as seen in exploratory and confirmatory factor analyses. We will use the short Hebrew version supplied by the questionnaire's authors.

Measure of attachment

Experiences in Close Relationships Scale (ECR), (Brennan et al., 1998). This measure examines patterns of attachment through a self-report questionnaire containing 36 items. The participants are required to rate to what extent each item describes his attitude toward close relationships, from (1) - strongly disagree, to (7) - strongly agree. 18 items relate to an insecure/anxious attachment pattern, and another 18 items relate to an insecure/avoidant attachment pattern. The original study reported Cronbach's alpha as .91 and .94 for the Anxiety and Avoidance subscales, respectively, and similar results have been found since (Vogel & Wei, 2005). Test-retest reliability has been shown to be around 0.7 (Lopez & Gormley, 2002). The Hebrew version of the questionnaire will be used in this study, translated by Mikulincer & Florian (2000). They also validated its two-factor structure on an Israeli sample, with high internal reliability (Cronbach's alpha .92 for anxious attachment and .93 for avoidant attachment).

Measure of emotion regulation The Differentiation of Self Inventory (DSI), (Skowron & Friedlander, 1998; Skowron & Schmitt, 2003). The DSI is a self-report questionnaire that measures self-other differentiation as well as adaptive emotional regulation, which are vital for the development of mentalizing ability. This is a self-report instrument for adults (age ≥25 years), that was modification translated to Hebrew and validated for adolescents and young adults (Rothschild-Yakar et al., 2016). We will use the Hebrew version of Skowron and Schmitt's (2003) revised edition comprising 46 items in four subscales (Emotional Reactivity, I Position, Emotional Cutoff and Fusion with Others). Participants rated items on a 6-point Likert-type response scale ranging from Not at all (1) to Very true (6). Higher scores indicate a greater level of differentiation. The DSI showed external validity, with elevated DSI scores predicting lower chronic anxiety and better psychological adjustment (Skowron & Friedlander, 1998). Internal consistency reliabilities of the DSI and its subscale calculated with Cronbach's alpha were reported as follows: DSI full scale=.88, Emotional Reactivity=.84, I Position=.83, Emotional Cutoff=.82, and Fusion with Others=.74 (Skowron & Friedlander, 1998).

Measures of background variables, comorbidity, and estimation of intellectual ability

Personal details questionnaire. This questionnaire covers basic personal details such as age, country of origin, formal education, past or present emotional difficulties, past or present symptoms of EDs and the height and weight of the participants, as well as family details such as parental marital status, socioeconomic status, and parental education.

The short Depression, Anxiety and Stress Scale (DASS)-21 - (Lovibond & Lovibond, 1995). The DASS-21 is a 21-item self-report measure designed to assess and discriminate between symptoms of depression, anxiety, and stress. It consists of 21 items, which participants rate on a scale of 0 to 3 about how accurately statements regarding depression, anxiety, and stress applied to them over the past week. The DASS-21 has demonstrated acceptable psychometric properties in clinical and nonclinical populations, with high internal consistency for each sub-scale ranging from α = .82 to .94 (Antony, Bieling, Cox, Enns, & Swinson, 1998; Henry & Crawford, 2005).

The Eating Attitudes Test (EAT-26): (Garner et al, 1982). The EAT-26 will be used to measure the presence and severity of EDs. This is a self-report questionnaire that examines the level of pathological eating-related preoccupations and behaviours. The EAT-26 includes three main subscales: (a) dieting, refraining from fatty food, and physical appearance; (b) bulimic symptomatology and preoccupation with food; and (c) personal control over eating habits. Participants rate the 26 items on a 6-point scale ranging from Never (1) to Always (6). High reliability and validity of the EAT-26 were found across different cultures (Garfinkel & Newman, 2001; Garner et al 1982), including in Israeli patients with EDs (Koslowsky et. al., 1992, Niv-Nadler, 1997).

The SCOFF- questionnaire for the assessment of eating disorders (Morgan et al., 1999). The SCOFF questionnaire is a simple 5- yes/no question tool, developed to screen for eating disorders in the general population. For every positive answer one point is given. A total score of two and above has been found to be 100% sensitive and 87.5% specific for the presence of any ED.

An estimated IQ: Similarities and block design subtests (Wechsler, 2008). Similarities and Block Design will be used as an estimate for IQ. The Similarities and Block Design subtests will be used from the Hebrew version of WAIS IIIHeb (Wechsler, 1997) for Adults. The two subtests were found to possess high loading on the factors to which they belong (Watkins et al, 2006).

Study procedure All tasks will be administrated individually by a master or doctoral student in a single two hours session. After receiving an information regarding the purpose of the study and its procedure the participants will sign a consent form. For participants under the age of 18, parental consent will be obtained as well. During the session the participants will complete online self-report questionnaires (personal details questionnaire, experiences in close relationships scale and the differentiation of self inventory) followed by the Hebrew version of the movie for assessment of social cognition (MASC-heb). Then the participants will complete an online self report questionnaire ( the Toronto alexithymia scale) followed by two computer tasks (the Cambridge mindreading face-voice battery and the reading the mind in the eyes),the Wechsler's Similarities and Block design and more online self- report questionnaires (the short depression, anxiety and stress scale, the reflective functioning questionnaire and the eating attitudes test 26).

To ascertain that the participants of the control group will not include participants suffering from EDs, they will pass the SCOFF questionnaire which is a common screening tool for Eds.

Control participants will be compensated for their participation by 80 NIS for their participation in the study. Control group sessions will take place in Haifa university.

20 participants (10 from the AN group and 10 from the control group) will be invited to a second half hour session, 2-6 month after the first session. The session will be administrated by a master or doctoral student. After receiving an information regarding the purpose of the study and its procedure the participants will sign a consent form. For participants under the age of 18, parental consent will be obtained as well. During the session the participant will complete the MASC-heb. Control participants will be compensated for their participation by 40 NIS for their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

• All patients will meet the DSM-5 (APA, 2013) criteria for diagnosis of AN on admission.

Exclusion Criteria:

• Patients will have no lifetime or current diagnosis of bipolar disorder, schizophrenia spectrum disorder, substance use disorder, mental retardation, organic brain syndrome, and any physical disorder except for inter-current medical problems.

Ages: 16 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — self identification
Study Population: Women hospitalized with AN at the ages 16-28.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Mentalization impairments measured by questionnaire | one year

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Ziv Hospital, Safed, Galilee
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No